CLINICAL TRIAL: NCT01407432
Title: Impact of Folates in the Care of the Male Infertility
Acronym: FOLFIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P 100108
Record Dates: First submitted 2011-06-28; First posted 2011-08-02 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-05

CONDITIONS: Male Infertility
Keywords: Male infertility; folic acid; in VITRO fertilization; sperm parameters; MTHFR genotype
MeSH Terms: conditions — Infertility, Male | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Folic acid (Experimental): tablets of 5 mg of folic acid
  Interventions: Drug: Folic acid
- Placebo (Placebo Comparator): Tablets of placebo of folic acid
  Interventions: Drug: placebo of folic acid

INTERVENTIONS:
Drug: Folic acid — Taking of folic acid 15 mg per day by hanging oral route during 3 at 4 months
  Arms: Folic acid
Drug: placebo of folic acid — Taking of placebo of folic acid by hanging oral route during 3 at 4 months
  Arms: Placebo

SUMMARY:
Unexplained male infertility is increasing, and, nowadays, the investigators only can propose palliative treatment, as In VITRO Fertilization (IVF). The folate metabolism is a key for the maintenance of genome integrity. A dysfunction in this pathway can be responsible of spermatogenesis defects, and further, of infertility. Few assays have shown that folate treatment can improve sperm parameters and fertility, till 30% in some of theses studies. The purpose of the investigators study is to demonstrate the impact of folates treatment on improvement of sperm parameters and on the rate of success of in VITRO fertilization procedures.

DETAILED DESCRIPTION:
The folate impact in the treatment of male infertility will be reviewed by this large multicentric randomized controlled double-blind study comparing 2 parallel groups of 184 patients. In each group: folic acid 15mg/day versus placebo, orally for at least 3 months (duration of a cycle of spermatogenesis). This assay will evaluate the effectiveness of treatment with folic acid compared to its placebo in infertile men with the outcome of IVF+/-ICSI techniques (pregnancy rate). It will also assess the impact of folate therapy on sperm parameters, and further, the impact on abnormal sperm DNA methylation profiles.

ELIGIBILITY:
Inclusion Criteria:

* Couple whose man is from 18 to 60 years old
* Couple whose man presents an infertility indicating a care in VITRO fertilization with or without intracytoplasmic sperm injection (IVF +/- ICSI)
* Couple whose spouse is from 18 to 38 years old
* Couple whose spouse do not present particular factors of infertility
* Couple Taken care in IVF +/- ICSI
* Couple with social insurance
* 2 members of the couple having signed the consent

Exclusion Criteria:

* Etiology of not genetic known male infertility : infertility of neoplastic origine, infertility of definitive obstructive origin
* Presence of a factor of feminine infertility : A definitive infertility tubal, Turned out ovarian incapacity (FSH > 9 and/or CFA <= 8)
* Male infertility requiring the appeal to some sperm testicular or in some frozen sperm- Men or women attend of HIV or hepatitis B or C
* Epileptic men
* Men under anti-folic treatment
* Men presenting a big sensibility to the folic acid or to one of the constituents of the drug
* Couple of which one of the partners refuses to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2011-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The rates of pregnancy in IVF +/- ICSI and spontaneous pregnancy according to the arm of treatment | 3 months
  Estimate the efficiency of the treatment by folic acid at infertile men on the improvement of improvement of the pregnancy rates in IVF +/- ICSI and spontaneous pregnancy before IVF +/- ICSI

SECONDARY OUTCOMES:
The rate of improvement of the sperm parameters with acid folic treatment | 3 months
  Estimate the efficiency of the treatment by folic acid on the sperm parameters
The rate of improvement of the nuclear quality of gametes with acid folic treatment | 3 months
  Estimate the efficiency of the treatment by folic acid on the nuclear quality of gametes
The rate of pregnancy of couple with infertile men treated by folic acid according to the methylene-tetrahydrofolate reductase (MTHFR) genotype | 3 months
  Estimate the impact of the methylene-tetrahydrofolate reductase (MTHFR) genotype of the patients on the rates of pregnancy according to the arm of treatment
The difference between the methylene-tetrahydrofolate reductase (MTHFR) genotype of the patients on sperm parameters according to the arm of treatment | 3 months
  Estimate the impact of methylene-tetrahydrofolate reductase (MTHFR) genotype of the patients on sperm parameters according to the arm of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle MATHIEU - D'ARGENT, MD, Principal Investigator — TENON Hospital - APHP
Locations (1):
- Service of gynaecology-obstetrics and medicine of the reproduction, Tenon Hospital - APHP, Paris, France

REFERENCES:
- [Background] Bentivoglio G, Melica F, Cristoforoni P. Folinic acid in the treatment of human male infertility. Fertil Steril. 1993 Oct;60(4):698-701. doi: 10.1016/s0015-0282(16)56225-6. PMID 8405528
- [Background] Bezold G, Lange M, Peter RU. Homozygous methylenetetrahydrofolate reductase C677T mutation and male infertility. N Engl J Med. 2001 Apr 12;344(15):1172-3. doi: 10.1056/NEJM200104123441517. No abstract available. PMID 11302150
- [Background] Blount BC, Mack MM, Wehr CM, MacGregor JT, Hiatt RA, Wang G, Wickramasinghe SN, Everson RB, Ames BN. Folate deficiency causes uracil misincorporation into human DNA and chromosome breakage: implications for cancer and neuronal damage. Proc Natl Acad Sci U S A. 1997 Apr 1;94(7):3290-5. doi: 10.1073/pnas.94.7.3290. PMID 9096386
- [Background] Boxmeer JC, Smit M, Weber RF, Lindemans J, Romijn JC, Eijkemans MJ, Macklon NS, Steegers-Theunissen RP. Seminal plasma cobalamin significantly correlates with sperm concentration in men undergoing IVF or ICSI procedures. J Androl. 2007 Jul-Aug;28(4):521-7. doi: 10.2164/jandrol.106.001982. Epub 2007 Feb 7. PMID 17287458
- [Background] Boxmeer JC, Macklon NS, Lindemans J, Beckers NG, Eijkemans MJ, Laven JS, Steegers EA, Steegers-Theunissen RP. IVF outcomes are associated with biomarkers of the homocysteine pathway in monofollicular fluid. Hum Reprod. 2009 May;24(5):1059-66. doi: 10.1093/humrep/dep009. Epub 2009 Feb 15. PMID 19221098
- [Background] Boxmeer JC, Smit M, Utomo E, Romijn JC, Eijkemans MJ, Lindemans J, Laven JS, Macklon NS, Steegers EA, Steegers-Theunissen RP. Low folate in seminal plasma is associated with increased sperm DNA damage. Fertil Steril. 2009 Aug;92(2):548-56. doi: 10.1016/j.fertnstert.2008.06.010. Epub 2008 Aug 22. PMID 18722602
- [Background] Chen J, Ma J, Stampfer MJ, Palomeque C, Selhub J, Hunter DJ. Linkage disequilibrium between the 677C>T and 1298A>C polymorphisms in human methylenetetrahydrofolate reductase gene and their contributions to risk of colorectal cancer. Pharmacogenetics. 2002 Jun;12(4):339-42. doi: 10.1097/00008571-200206000-00011. PMID 12042673
- [Background] Choi SW, Mason JB. Folate and colorectal carcinogenesis: is DNA repair the missing link? Am J Gastroenterol. 1998 Nov;93(11):2013-6. doi: 10.1111/j.1572-0241.1998.02013.x. No abstract available. PMID 9820367
- [Background] Doerksen T, Benoit G, Trasler JM. Deoxyribonucleic acid hypomethylation of male germ cells by mitotic and meiotic exposure to 5-azacytidine is associated with altered testicular histology. Endocrinology. 2000 Sep;141(9):3235-44. doi: 10.1210/endo.141.9.7661. PMID 10965894
- [Background] Ebisch IM, van Heerde WL, Thomas CM, van der Put N, Wong WY, Steegers-Theunissen RP. C677T methylenetetrahydrofolate reductase polymorphism interferes with the effects of folic acid and zinc sulfate on sperm concentration. Fertil Steril. 2003 Nov;80(5):1190-4. doi: 10.1016/s0015-0282(03)02157-5. PMID 14607573
- [Background] Eskenazi B, Kidd SA, Marks AR, Sloter E, Block G, Wyrobek AJ. Antioxidant intake is associated with semen quality in healthy men. Hum Reprod. 2005 Apr;20(4):1006-12. doi: 10.1093/humrep/deh725. Epub 2005 Jan 21. PMID 15665024
- [Background] Goyette P, Sumner JS, Milos R, Duncan AM, Rosenblatt DS, Matthews RG, Rozen R. Human methylenetetrahydrofolate reductase: isolation of cDNA mapping and mutation identification. Nat Genet. 1994 Aug;7(4):551. No abstract available. PMID 7951330
- [Background] Heijmans BT, Gussekloo J, Kluft C, Droog S, Lagaay AM, Knook DL, Westendorp RG, Slagboom EP. Mortality risk in men is associated with a common mutation in the methylene-tetrahydrofolate reductase gene (MTHFR). Eur J Hum Genet. 1999 Feb-Mar;7(2):197-204. doi: 10.1038/sj.ejhg.5200283. PMID 10196703
- [Background] Kelly TL, Li E, Trasler JM. 5-aza-2'-deoxycytidine induces alterations in murine spermatogenesis and pregnancy outcome. J Androl. 2003 Nov-Dec;24(6):822-30. doi: 10.1002/j.1939-4640.2003.tb03133.x. PMID 14581508
- [Background] Kelly TL, Neaga OR, Schwahn BC, Rozen R, Trasler JM. Infertility in 5,10-methylenetetrahydrofolate reductase (MTHFR)-deficient male mice is partially alleviated by lifetime dietary betaine supplementation. Biol Reprod. 2005 Mar;72(3):667-77. doi: 10.1095/biolreprod.104.035238. Epub 2004 Nov 17. PMID 15548731
- [Background] Kim YI, Pogribny IP, Basnakian AG, Miller JW, Selhub J, James SJ, Mason JB. Folate deficiency in rats induces DNA strand breaks and hypomethylation within the p53 tumor suppressor gene. Am J Clin Nutr. 1997 Jan;65(1):46-52. doi: 10.1093/ajcn/65.1.46. PMID 8988912
- [Background] Koury MJ, Horne DW, Brown ZA, Pietenpol JA, Blount BC, Ames BN, Hard R, Koury ST. Apoptosis of late-stage erythroblasts in megaloblastic anemia: association with DNA damage and macrocyte production. Blood. 1997 Jun 15;89(12):4617-23. PMID 9192787
- [Background] Kundu TK, Rao MR. CpG islands in chromatin organization and gene expression. J Biochem. 1999 Feb;125(2):217-22. doi: 10.1093/oxfordjournals.jbchem.a022276. PMID 9990116
- [Background] Lengauer C, Kinzler KW, Vogelstein B. DNA methylation and genetic instability in colorectal cancer cells. Proc Natl Acad Sci U S A. 1997 Mar 18;94(6):2545-50. doi: 10.1073/pnas.94.6.2545. PMID 9122232
- [Background] Ma J, Stampfer MJ, Giovannucci E, Artigas C, Hunter DJ, Fuchs C, Willett WC, Selhub J, Hennekens CH, Rozen R. Methylenetetrahydrofolate reductase polymorphism, dietary interactions, and risk of colorectal cancer. Cancer Res. 1997 Mar 15;57(6):1098-102. PMID 9067278
- [Background] Matsushita S, Muramatsu T, Arai H, Matsui T, Higuchi S. The frequency of the methylenetetrahydrofolate reductase-gene mutation varies with age in the normal population. Am J Hum Genet. 1997 Dec;61(6):1459-60. doi: 10.1086/301640. No abstract available. PMID 9399898
- [Background] Oliva A, Dotta A, Multigner L. Pentoxifylline and antioxidants improve sperm quality in male patients with varicocele. Fertil Steril. 2009 Apr;91(4 Suppl):1536-9. doi: 10.1016/j.fertnstert.2008.09.024. Epub 2008 Nov 5. PMID 18990381
- [Background] Ravel C, Chantot-Bastaraud S, Chalmey C, Barreiro L, Aknin-Seifer I, Pfeffer J, Berthaut I, Mathieu EE, Mandelbaum J, Siffroi JP, McElreavey K, Bashamboo A. Lack of association between genetic polymorphisms in enzymes associated with folate metabolism and unexplained reduced sperm counts. PLoS One. 2009 Aug 6;4(8):e6540. doi: 10.1371/journal.pone.0006540. PMID 19657388
- [Background] Rosenberg N, Murata M, Ikeda Y, Opare-Sem O, Zivelin A, Geffen E, Seligsohn U. The frequent 5,10-methylenetetrahydrofolate reductase C677T polymorphism is associated with a common haplotype in whites, Japanese, and Africans. Am J Hum Genet. 2002 Mar;70(3):758-62. doi: 10.1086/338932. Epub 2002 Jan 4. PMID 11781870
- [Background] Rozen R, Fraser FC, Shaw G. Decreased proportion of female newborn infants homozygous for the 677 C-->T mutation in methylenetetrahydrofolate reductase. Am J Med Genet. 1999 Mar 12;83(2):142-3. doi: 10.1002/(sici)1096-8628(19990312)83:23.0.co;2-y. No abstract available. PMID 10190487
- [Background] Skjelbred CF, Svendsen M, Haugan V, Eek AK, Clausen KO, Svendsen MV, Hansteen IL. Influence of DNA repair gene polymorphisms of hOGG1, XRCC1, XRCC3, ERCC2 and the folate metabolism gene MTHFR on chromosomal aberration frequencies. Mutat Res. 2006 Dec 1;602(1-2):151-62. doi: 10.1016/j.mrfmmm.2006.08.009. Epub 2006 Sep 25. PMID 16997330
- [Background] Stegmann K, Ziegler A, Ngo ET, Kohlschmidt N, Schroter B, Ermert A, Koch MC. Linkage disequilibrium of MTHFR genotypes 677C/T-1298A/C in the German population and association studies in probands with neural tube defects(NTD). Am J Med Genet. 1999 Nov 5;87(1):23-9. PMID 10528242
- [Background] Szymanski W, Kazdepka-Zieminska A. [Effect of homocysteine concentration in follicular fluid on a degree of oocyte maturity]. Ginekol Pol. 2003 Oct;74(10):1392-6. Polish. PMID 14669450
- [Background] Wong WY, Merkus HM, Thomas CM, Menkveld R, Zielhuis GA, Steegers-Theunissen RP. Effects of folic acid and zinc sulfate on male factor subfertility: a double-blind, randomized, placebo-controlled trial. Fertil Steril. 2002 Mar;77(3):491-8. doi: 10.1016/s0015-0282(01)03229-0. PMID 11872201
- [Derived] de Ligny W, Smits RM, Mackenzie-Proctor R, Jordan V, Fleischer K, de Bruin JP, Showell MG. Antioxidants for male subfertility. Cochrane Database Syst Rev. 2022 May 4;5(5):CD007411. doi: 10.1002/14651858.CD007411.pub5. PMID 35506389